CLINICAL TRIAL: NCT02338960
Title: Phase 3, Randomized, Double-blind, Placebo-controlled, Trial With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Subcutaneously Bremelanotide in Premenopausal Women With Hypoactive Sexual Desire Disorder (HSDD)
Brief Title: 2. Study to Evaluate the Efficacy/Safety of Bremelanotide in Premenopausal Women With Hypoactive Sexual Desire Disorder
Acronym: HSDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMT-302; Reconnect Study (Other: Palatin Technologies)
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-12

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD Female; Sexual Desire Disorder; decreased desire; female sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bremelanotide (BMT/BMT) (Experimental): (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  (OLE Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Interventions: Drug: Bremelanotide
- Placebo (PBO/BMT) (Placebo Comparator): (Main Study) PBO administered SC on an as-desired basis for 24 weeks
  (OLE Study) subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Interventions: Drug: Bremelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Bremelanotide — A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
  Other Names: BMT; PT-141
Drug: Placebo — Placebo
  Other Names: PBO
  Arms: Placebo (PBO/BMT)

SUMMARY:
A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial with an optional Open-label Extension to evaluate the efficacy of bremelanotide (BMT), administered subcutaneously (SC) on an as needed basis for the treatment of HSDD (with or without decreased arousal) in premenopausal females.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, placebo-controlled, parallel group study in up to 80 sites in the United States of America (USA) and Canada to evaluate the efficacy and safety of a fixed dose of SC BMT versus placebo on an as-needed basis under conditions of home use in premenopausal women with HSDD (with or without decreased arousal).

The study will consist of 2 phases: (1) Core Study: 4-week no-treatment qualification period, a 4-week single-blind placebo treatment period (baseline), and a 24-week double-blind treatment period where participants will self-administer placebo or BMT 1.75 mg SC via an autoinjector; and (2) Extension Phase: a 52-week open-label treatment period during which all subjects will receive BMT 1.75 mg.

Primary Objective

• To evaluate the efficacy of bremelanotide (BMT), administered subcutaneously (SC) on an as needed basis for the treatment of HSDD (with or without decreased arousal) in premenopausal females.

Secondary Objectives

* To evaluate the efficacy of BMT in premenopausal women in the double-blind Core Study, as assessed by subject responses to questionnaires measuring sexual function, treatment satisfaction, and distress associated with sexual dysfunction.
* To evaluate the safety of BMT in premenopausal women in the double-blind Core Study.
* To evaluate the safety of long-term therapy with BMT in the open label Extension Phase.
* To evaluate the efficacy of long-term therapy with BMT in the open-label Extension Phase.

ELIGIBILITY:
Main Inclusion Criteria:

* Has met diagnostic criteria for HSDD for at least 6 months
* Is willing and able to understand and comply with all study requirements
* Has a normal pelvic examination at screening

Main Exclusion Criteria:

* Subjects should be generally healthy premenopausal females with no psychological, gynecological or urological conditions which might contribute to the sexual dysfunction, compromise study participation, or confound interpretation of the study results
* Not currently under treatment for the sexual dysfunction and willing to forego other treatments through the course of the clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jordan, Study Director — Palatin Technologies, Inc
Locations (91):
- United States (87):
  - Palatin Clinical Site 242, Birmingham, Alabama
  - Palatin Clinical Site 218, Phoenix, Arizona
  - Palatin Clinical Site 254, Tucson, Arizona
  - Palatin Clinical Site 207, Hot Springs, Arkansas
  - Palatin Clinical Site 258, Beverly Hills, California
  - Palatin Clinical Site 256, Garden Grove, California
  - Palatin Clinical Site 291, Los Angeles, California
  - Palatin Clinical Site 270, Oakland, California
  - Palatin Clinical Site 210, San Diego, California
  - Palatin Clinical Site 251, San Diego, California
  - Palatin Clinical Site 272, Sherman Oaks, California
  - Palatin Clinical Site 253, Tarzana, California
  - Palatin Clinical Site 212, Denver, Colorado
  - Palatin Clinical Site 219, Denver, Colorado
  - Palatin Clinical Site 243, Lakewood, Colorado
  - Palatin Clinical Site 211, New London, Connecticut
  - Palatin Clinical Site 229, Waterbury, Connecticut
  - Palatin Clinical Site 202, Washington D.C., District of Columbia
  - Palatin Clinical Site 204, Aventura, Florida
  - Palatin Clinical Site 273, Coral Gables, Florida
  - Palatin Clinical Site 203, Fort Myers, Florida
  - Palatin Clinical Site 255, Gainesville, Florida
  - Palatin Clinical Site 266, Gainesville, Florida
  - Palatin Clinical Site 224, Jupiter, Florida
  - Palatin Clinical Site 250, Orlando, Florida
  - Palatin Clinical Site 261, Oviedo, Florida
  - Palatin Clinical Site 260, Pinellas Park, Florida
  - Palatin Clinical Site 236, West Palm Beach, Florida
  - Palatin Clinical Site 248, Alpharetta, Georgia
  - Palatin Clinical Site 263, Atlanta, Georgia
  - Palatin Clinical Site 288, Addison, Illinois
  - Palatin Clinical Site 252, Chicago, Illinois
  - Palatin Clinical Site 201, Chicago, Illinois
  - Palatin Clinical Site 277, Indianapolis, Indiana
  - Palatin Clinical Site 247, Prairie Village, Kansas
  - Palatin Clinical Site 286, Paducah, Kentucky
  - Palatin Clinical Site 279, Lake Charles, Louisiana
  - Palatin Clinical Site 281, Metairie, Louisiana
  - Palatin Clinical Site 257, Annapolis, Maryland
  - Palatin Clinical Site 222, Lutherville, Maryland
  - Palatin Clinical Site 283, Rockville, Maryland
  - Palatin Clinical Site 265, Boston, Massachusetts
  - Palatin Clinical Site 217, New Bedford, Massachusetts
  - Palatin Clinical Site 239, Kalamazoo, Michigan
  - Palatin Clinical Site 245, Saginaw, Michigan
  - Palatin Clinical Site 287, Flowood, Mississippi
  - Palatin Clinical Site 244, Kansas City, Missouri
  - Palatin Clinical Site 280, St Louis, Missouri
  - Palatin Clinical Site 220, Lincoln, Nebraska
  - Palatin Clinical Site 290, Berlin, New Jersey
  - Palatin Clinical Site 233, Lawrenceville, New Jersey
  - Palatin Clinical Site 276, Albuquerque, New Mexico
  - Palatin Clinical Site 282, Rochester, New York
  - Palatin Clinical Site 264, Cary, North Carolina
  - Palatin Clinical Site 206, Raleigh, North Carolina
  - Palatin Clinical Site 231, Salisbury, North Carolina
  - Palatin Clinical Site 209, Winston-Salem, North Carolina
  - Palatin Clinical Site 271, Canton, Ohio
  - Palatin Clinical Site 215, Cincinnati, Ohio
  - Palatin Clinical Site 232, Cleveland, Ohio
  - Palatin Clinical Site 246, Columbus, Ohio
  - Palatin Clinical Site 221, Mayfield Heights, Ohio
  - Palatin Clinical Site 289, Tiffin, Ohio
  - Palatin Clinical Site 238, Oklahoma City, Oklahoma
  - Palatin Clinical Site 227, Oklahoma City, Oklahoma
  - Palatin Clinical Site 267, Allentown, Pennsylvania
  - Palatin Clinical Site 234, Philadelphia, Pennsylvania
  - Palatin Clinical Site 240, Pittsburgh, Pennsylvania
  - Palatin Clinical Site 278, Lincoln, Rhode Island
  - Palatin Clinical Site 200, Greer, South Carolina
  - Palatin Clinical Site 259, Moncks Corner, South Carolina
  - Palatin Clinical Site 275, Chattanooga, Tennessee
  - Palatin Clinical Site 216, Jackson, Tennessee
  - Palatin Clinical Site 274, Memphis, Tennessee
  - Palatin Clinical Site 292, Nashville, Tennessee
  - Palatin Clinical Site 235, Arlington, Texas
  - Palatin Clinical Site 230, Austin, Texas
  - Palatin Clinical Site 223, Dallas, Texas
  - Palatin Clinical Site 208, Houston, Texas
  - Palatin Clinical Site 269, Draper, Utah
  - Palatin Clinical Site 228, West Jordan, Utah
  - Palatin Clinical Site 284, Newport News, Virginia
  - Palatin Clinical Site 205, Norfolk, Virginia
  - Palatin Clinical Site 213, Richmond, Virginia
  - Palatin Clinical Site 268, Richmond, Virginia
  - Palatin Clinical Site 214, Seattle, Washington
  - Palatin Clinical Site 285, Charleston, West Virginia
- Canada (4):
  - Palatin Clinical Site 400, Vancouver, British Columbia
  - Palatin Clinical Site 405, Greater Sudbury, Ontario
  - Palatin Clinical Site 401, Pointe-Claire, Quebec
  - Palatin Clinical Site 404, Sherbrooke, Quebec

REFERENCES:
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Derived] Spielmans GI, Ellefson EM. Small Effects, Questionable Outcomes: Bremelanotide for Hypoactive Sexual Desire Disorder. J Sex Res. 2024 May;61(4):540-561. doi: 10.1080/00224499.2023.2175192. Epub 2023 Feb 21. PMID 36809187
- [Derived] Clayton AH, Kingsberg SA, Portman D, Sadiq A, Krop J, Jordan R, Lucas J, Simon JA. Safety Profile of Bremelanotide Across the Clinical Development Program. J Womens Health (Larchmt). 2022 Feb;31(2):171-182. doi: 10.1089/jwh.2021.0191. PMID 35147466
- [Derived] Koochaki P, Revicki D, Wilson H, Pokrzywinski R, Jordan R, Lucas J, Williams LA, Sadiq A, Krop J. The Patient Experience of Premenopausal Women Treated with Bremelanotide for Hypoactive Sexual Desire Disorder: RECONNECT Exit Study Results. J Womens Health (Larchmt). 2021 Apr;30(4):587-595. doi: 10.1089/jwh.2020.8460. Epub 2021 Feb 3. PMID 33538638
- [Derived] Revicki DA, Althof SE, Derogatis LR, Kingsberg SA, Wilson H, Sadiq A, Krop J, Jordan R, Lucas J. Reliability and validity of the elements of desire questionnaire in premenopausal women with hypoactive sexual desire disorder. J Patient Rep Outcomes. 2020 Oct 8;4(1):82. doi: 10.1186/s41687-020-00241-6. PMID 33033885
- [Derived] Simon JA, Kingsberg SA, Portman D, Williams LA, Krop J, Jordan R, Lucas J, Clayton AH. Long-Term Safety and Efficacy of Bremelanotide for Hypoactive Sexual Desire Disorder. Obstet Gynecol. 2019 Nov;134(5):909-917. doi: 10.1097/AOG.0000000000003514. PMID 31599847
- [Derived] Kingsberg SA, Clayton AH, Portman D, Williams LA, Krop J, Jordan R, Lucas J, Simon JA. Bremelanotide for the Treatment of Hypoactive Sexual Desire Disorder: Two Randomized Phase 3 Trials. Obstet Gynecol. 2019 Nov;134(5):899-908. doi: 10.1097/AOG.0000000000003500. PMID 31599840
- [Derived] Clayton AH, Lucas J, DeRogatis LR, Jordan R. Phase I Randomized Placebo-controlled, Double-blind Study of the Safety and Tolerability of Bremelanotide Coadministered With Ethanol in Healthy Male and Female Participants. Clin Ther. 2017 Mar;39(3):514-526.e14. doi: 10.1016/j.clinthera.2017.01.018. Epub 2017 Feb 9. PMID 28189361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Core ("Main") Study consisted of a 4-week no drug Screening period, followed by a 4-week single blind PBO period, first dose administered in-clinic. Following the end of single-blind period, which served as Baseline, eligible subjects were then randomized to a 24-week double-blind outpatient treatment period, first dose administered in-clinic.
Pre-assignment Details: Core Study: 703 participants enrolled, 89 run-in failures 614 participants were randomized.
  OLE Study (optional): Of the 392 completers of the Core study, 321 participants enrolled in optional OLE study. The OLE Study was not reported.
Groups:
- Placebo PBO/BMT: Core Study: Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks.
  Placebo
  OLE Study: Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Brememlanotide BMT/BMT: Core and OLE Study: Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Period: Core Study
Arm/Group | Placebo PBO/BMT | Brememlanotide BMT/BMT
Started | 306 | 308
Received Intervention | 303 | 301
Completed | 219 | 173
Not Completed | 87 | 135
Period: Open Label Extension
Arm/Group | Placebo PBO/BMT | Brememlanotide BMT/BMT
Started (321/392 Subjects who completed the Core Study continued into the optional OLE study.) | 191 | 130
Completed | 77 | 51
Not Completed | 114 | 79

BASELINE CHARACTERISTICS:
Population: Randomized population = 614, of which 10 were not dosed, leaving 604 participants. A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 130 in the BMT group (BMT-BMT) and 191 in the PBO group (PBO-BMT)
Groups:
- Bremelanotide (BMT/BMT): Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours (Main) followed by a 52-week open label extension study (OLE)
  BMT/BMT
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo (PBO/BMT): Subjects will self-administer a fixed dose of placebo (PBO) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours (Main) followed by a 52-week open label extension study (OLE) where participants receive only BMT, no placebo
  PBO/BMT
  Placebo: Placebo bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Total: Total of all reporting groups
Arm/Group | Bremelanotide (BMT/BMT) | Placebo (PBO/BMT) | Total
Number analyzed (Participants) | 303 | 301 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into OLE Study Phase, including 130 in the BMT group (BMT/BMT) and 191 in the PBO group (PBO/BMT).
  years
    Main | 38.5 (7.19) | 39.1 (6.96) | 38.8 (7.08)
    OLE: number analyzed (Participants) | 130 | 191 | 321
    OLE | 39.8 (7.12) | 39.4 (6.54) | 39.6 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into OLE Study Phase, including 130 in the BMT group (BMT/BMT) and 191 in the PBO group (PBO/BMT).
  Participants
    Main: Female | 303 | 301 | 604
    Main: Male | 0 | 0 | 0
    OLE: number analyzed (Participants) | 130 | 191 | 321
    OLE: Female | 130 | 191 | 321
    OLE: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into OLE Study Phase, including 130 in the BMT group (BMT/BMT) and 191 in the PBO group (PBO/BMT).
  Participants
    Main: Hispanic or Latino | 21 | 21 | 42
    Main: Not Hispanic or Latino | 282 | 280 | 562
    Main: Unknown or Not Reported | 0 | 0 | 0
    OLE: number analyzed (Participants) | 130 | 191 | 321
    OLE: Hispanic or Latino | 6 | 9 | 15
    OLE: Not Hispanic or Latino | 124 | 182 | 306
    OLE: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into OLE Study Phase, including 130 in the BMT group (BMT/BMT) and 191 in the PBO group (PBO/BMT).
  Participants
    Main: American Indian or Alaska Native | 2 | 1 | 3
    Main: Asian | 5 | 4 | 9
    Main: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Main: Black or African American | 29 | 29 | 58
    Main: White | 263 | 262 | 525
    Main: More than one race | 3 | 2 | 5
    Main: Unknown or Not Reported | 1 | 3 | 4
    OLE: number analyzed (Participants) | 130 | 191 | 321
    OLE: American Indian or Alaska Native | 0 | 0 | 0
    OLE: Asian | 1 | 2 | 3
    OLE: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    OLE: Black or African American | 10 | 15 | 25
    OLE: White | 117 | 171 | 288
    OLE: More than one race | 2 | 2 | 4
    OLE: Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of a Fixed Dose of Bremelanotide as Measured by FSFI (Question Q1 and Q2), 28-day Recall.
Description: As measured by change from baseline to end-of-study in the desire domain from the FSFI (Question Q1 and Q2), 28-day recall, co-primary endpoint - FSFI desire domain
  This score is on a scale ranging from 1.2 to 6. A higher score on this scale represent an increase in sexual desire and is a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bremelanotide BMT/BMT: (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  (OLE Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo PBO/BMT: (Main Study) PBO administered SC on an as-desired basis for 24 weeks
  Placebo: Placebo
  (OLE Study) subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 288
score on a scale
  Main study | 0.63 (1.036) | 0.21 (0.922)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | 1.25 (1.158) | 0.70 (1.220)

2. Primary Outcome: Efficacy of a Fixed Dose of Bremelanotide as Measured by FSDS-DAO (Item 13)
Description: As measured by the change from baseline to End-of-Study of the Core Study in the bothered by low desire item from the FSDS-DAO (item 13).
  Responses range from 0 (never) to 4 (always). Lower scores on this scale represent an increase in sexual desire and indicate a better outcome.
  Higher scores indicate a worse outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 288
score on a scale
  Main study: number analyzed (Participants) | 282 | 285
  Main study | -0.71 (1.145) | -0.42 (1.047)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | -1.4 (1.20) | -0.9 (1.07)

3. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study (EOS) in the Number of Satisfying Sexual Events (SSEs) Associated With Study Drug Administration
Description: Mean change from Baseline to end of study (EOS) in the number of satisfying sexual events (SSEs) that occurred within 16 hours of study drug dosing and reported within 72 hours. An increase in number indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total 321 of the 392 (81.9%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase. 128 participants in the OLE study completed the 52 weeks.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
events
  Main study | 0.0 (1.34) | 0.0 (1.20)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.19 (1.997) | -0.31 (1.296)

4. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in Mean Desire Score (Q3) From the FSEP-R
Description: FSEP-R=Female Sexual Encounter Profile - Revised Scores on this scale range from 0 (no desire) to 3 (high desire). Scale is derived from a questionnaire (mean desire score) where an increase in value indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
score on a scale
  Main study | 0.04 (1.065) | 0.01 (0.928)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.43 (1.095) | 0.33 (1.023)

5. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in Mean Satisfaction With Desire Score (Q4) From FSEP-R
Description: FSEP-R=Female Sexual Encounter Profile - Revised Scores range from 0 (no desire) to 3 (high desire). Scale is derived from a questionnaire (mean desire score) where a higher score indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
score on a scale
  Main study | 0.27 (1.077) | 0.11 (0.977)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.76 (1.127) | 0.47 (1.075)

6. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the FSDS-DAO Total Score
Description: FSDS-DAO = Female Sexual Distress Scale - Desire/Arousal/Orgasm. The FSDS-DAO is a validated 15-item self-assessment of sexual feelings and problems. All responses are on a scale ranging from 0 ("never") to 4 ("always").
  Total Scores range from 0 (never feel bothered) to 60 (always feel bothered). Decreased scores indicate improvement. A higher score on this scale indicates a worse outcome. The score is the mean change from Baseline observed at EOS (Baseline score - EOS score)
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 285
score on a scale
  Main study | -9.7 (13.79) | -5.6 (12.06)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | -18.4 (14.06) | -11.1 (14.37)

7. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the FSFI Total Score
Description: Female Sexual Function Index (FSFI) The score is computed programmatically ] resulting in a score on a scale ranging from 1.2 to 6 (Note: OLE: Open-label extension. Scores range from 2 to 36. An improvement in total FSFI score is an increase from baseline. A higher score on this scale represents an increase in sexual desire and is a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 288
score on a scale
  Main study | 2.45 (7.383) | 0.84 (5.879)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | 5.15 (7.301) | 3.14 (7.281)

8. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Mean Level of Sexual Arousal (Q6) From the FSEP-R
Description: FSEP-R=Female Sexual Encounter Profile - Revised Scores on this scale range from 0 (no desire) to 3 (high desire) Scale is derived from a questionnaire (mean desire score) where a higher score indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
score on a scale
  Main study | 0.04 (1.068) | -0.01 (0.906)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.33 (0.987) | 0.35 (0.994)

9. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Mean Satisfaction With Sexual Arousal (Q7) From the FSEP-R
Description: FSEP-R=Female Sexual Encounter Profile - Revised Scores range from 0 (no desire) to 3 (high desire) Scale is derived from a questionnaire (mean desire score) where a higher score indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
score on a scale
  Main study | 0.23 (1.112) | 0.09 (0.974)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.60 (1.107) | 0.47 (1.102)

10. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Scored Time Spent Being Concerned by Difficulty With Sexual Arousal (Q14) From the FSDS-DAO
Description: FSDS-DAO = Female Sexual Distress Scale - Desire/Arousal/Orgasm.
  The FSDS-DAO is a validated 15-item self-assessment of sexual feelings and problems. Scores on this scale range from 0 ("never") to 4 ("always"). Decreased scores indicate improvement.
  A higher score on this scale indicates a worse outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 285
score on a scale
  Main study | -0.8 (1.23) | -0.4 (1.11)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | -1.3 (1.11) | -0.9 (1.17)

11. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Arousal Domain of the FSFI (Q3 to Q6)
Description: Female Sexual Function Index (FSFI)
  The score is computed programmatically using the algorithm described by Rosen, resulting in a score ranging from 1.2 to 6. Higher scores on this scale represent an increase in sexual desire and is a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 288
score on a scale
  Main study | 0.52 (1.535) | 0.18 (1.254)
  Open label extension: number analyzed (Participants) | 53 | 75
  Open label extension | 1.19 (1.560) | 0.83 (1.563)

12. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Total Number of SSEs
Description: Change from Baseline to EOS in the total number of satisfying sexual events SSEs. A higher number of events indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 282 | 290
events
  Main study | 0.0 (1.34) | -0.0 (1.20)
  Open label extension: number analyzed (Participants) | 53 | 80
  Open label extension | 0.25 (2.376) | -0.35 (1.655)

13. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Desire Domain of the FSFI (Q1 to Q2) Throughout the Entirety of the Double-blind Phase
Description: FSFI = Female Sexual Function Index
  The score is on a scale ranging from 1.2 to 6. A higher score on this scale represents an increase in sexual desire and is a better outcome.
Time Frame: 24 weeks (Main Study)
Population: Completed double-blind study of Main study. OLE study was not a double blind study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bremelanotide BMT: (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo PBO: Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Placebo: Placebo
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 173 | 219
score on a scale | 0.78 (1.052) | 0.16 (0.909)

14. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Score for Feeling Bothered by Low Sexual Desire as Measured by the FSDS-DAO (Item 13) Throughout the Entirety of the Double-blind Phase
Description: FSDS-DAO = Female Sexual Distress Scale - Desire/Arousal/Orgasm.
  The FSDS-DAO is a validated 15-item self-assessment of sexual feelings and problems. The score is on a scale ranging from 0 ("never") to 4 ("always"). Decreased scores indicate improvement. A higher score indicates a worse outcome.
Time Frame: 24 weeks (Main Study)
Population: Completed double-blind study of Main study. OLE study wan not a double blind study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bremelanotide BMT: (Main Study) Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 173 | 218
score on a scale | -0.8 (1.22) | -0.4 (1.02)

15. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Number of SSEs Associated With Study Drug Administration Throughout the Entirety of the Double-blind Phase
Description: Mean change from Baseline to EOS in the number of satisfying sexual events SSEs associated with study drug administration throughout the entirety of the double-blind phase. A higher number of events indicates a better outcome.
Time Frame: 24 weeks (Main Study)
Population: Completed double-blind study of Main study. OLE study wan not a double blind study.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 177 | 221
events | 0.1 (1.37) | -0.1 (1.28)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Reporting participants: all subjects who were randomized and used at least 1 dose of double-blind study drug.
Groups:
- Bremelanotide (Main Study); Bremelanotide (OLE); Placebo (OLE): Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo (Main Study): Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Placebo: Placebo
Arm/Group | Bremelanotide (Main Study) | Placebo (Main Study) | Bremelanotide (OLE) | Placebo (OLE)
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/301 | 0/130 | 0/191
Serious Adverse Events (participants affected / at risk) | 3/303 | 2/301 | 1/130 | 0/191
Other Adverse Events (participants affected / at risk) | 224/303 | 137/301 | 93/130 | 142/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bremelanotide (Main Study) (N=303) | Placebo (Main Study) (N=301) | Bremelanotide (OLE) (N=130) | Placebo (OLE) (N=191)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bremelanotide (Main Study) (N=303) | Placebo (Main Study) (N=301) | Bremelanotide (OLE) (N=130) | Placebo (OLE) (N=191)
Nausea (Gastrointestinal disorders) | 111 | 0 | 37 | 84
Vomiting (Gastrointestinal disorders) | 13 | 1 | 3 | 9
Sinusitis (Infections and infestations) | 14 | 13 | 4 | 9
Upper respiratory tract infection (Infections and infestations) | 12 | 13 | 5 | 7
Urinary tract infection (Infections and infestations) | 10 | 9 | 4 | 11
Nasopharyngitis (Infections and infestations) | 9 | 18 | 4 | 10
Injection site pain (General disorders) | 21 | 17 | 2 | 5
Injection site reaction (General disorders) | 16 | 0 | 4 | 5
Injection site erythema (General disorders) | 10 | 0 | 2 | 3
Fatigue (General disorders) | 8 | 2 | 3 | 5
Injection site hematoma (General disorders) | 7 | 4 | 0 | 4
Headache (Nervous system disorders) | 38 | 4 | 9 | 29
Paresthesia (Nervous system disorders) | 9 | 0 | 1 | 4
Flushing (Vascular disorders) | 43 | 0 | 11 | 41
Hot flush (Vascular disorders) | 11 | 0 | 0 | 8
Sunburn (Injury, poisoning and procedural complications) | 16 | 28 | 22 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 1 | 5
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 4 | 1
Bronchitis (Infections and infestations) | 5 | 4 | 4 | 2
Fungal infection (Infections and infestations) | 4 | 4 | 2 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 5 | 5 | 0 | 6
Dizziness (Nervous system disorders) | 4 | 2 | 0 | 5
Migraine (Nervous system disorders) | 0 | 2 | 3 | 2
Influenza like illness (General disorders) | 2 | 0 | 2 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4
Blood creatine phophokinase (Investigations) | 4 | 0 | 0 | 4
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 4
Depression (Psychiatric disorders) | 0 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.